CLINICAL TRIAL: NCT03844568
Title: Nocturnal Nasal Continuous Positive Airway Pressure in Aspiration Pneumonia
Acronym: NAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Hard to recruit due to COVID-19 issue.
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Eun Sun Kim, Associate professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1809-493-002
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Aspiration Pneumonia
Keywords: aspiration pneumonia; continuous positive airway pressure, CPAP
MeSH Terms: conditions — Pneumonia, Aspiration; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal CPAP group (Experimental): Applying nocturnal nasal continuous positive airway pressure in additional to usual pneumonia treatment
  Interventions: Device: nocturnal nasal continuous positive airway pressure
- Control group (No Intervention): Usual pneumonia treatment

INTERVENTIONS:
Device: nocturnal nasal continuous positive airway pressure — applying nasal continuous positive airway pressure at 7.5-10cmH2O for at least 4 hours during nighttime
  Arms: nasal CPAP group

SUMMARY:
Numerous elderly patients are suffering from aspiration pneumonia due to anatomical or functional predisposing factors including enteral tube feeding, swallowing difficulties, and gastroesophageal reflux disease (GERD). Previous studies have been demonstrated that continuous positive airway pressure (CPAP) is an acceptable means of managing chronic aspiration, atelectasis, and GERD. The purpose of this study is to determine whether nocturnal nasal CPAP is beneficial in patients with aspiration pneumonia and that it would contribute to the rapid clinical stability of aspiration pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Diagnosis of pneumonia: the presence of new pulmonary infiltration in dependent areas on chest radiographs at the time of hospitalization with at least one of the following

  1. New or increased cough
  2. Abnormal temperature (< 35.6℃ or > 37.8℃)
  3. Abnormal serum leukocyte count (leukocytosis, left shift, or leukopenia)
* Aspiration tendency or risk factors for frequent or large volume aspiration with at least one of the following

  1. Altered mental status
  2. Gastrointestinal disorder
  3. Dysphagia or swallowing difficulties
  4. Esophageal motility disorders
  5. Tracheostomy state
  6. Enteral tube feeding
* Informed consent

Exclusion Criteria:

* Severe hypercapnia (PaCO2 > 70mmHg)
* Respiratory arrest requiring tracheal intubation
* Cardiac arrest, acute coronary syndrome or life threatening arrhythmias
* Failure of more than two organs
* Recent trauma or burns of the neck and face
* Non- cooperation
* Pregnancy
* Withdrawal of consent
* Refusal of treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Time to clinical stability-respiration (CS-r) | up to 2 weeks
  time to respiratory stabilization (respiratory rate ≤ 24/min and arterial oxygen saturation ≥ 90% or a partial pressure of oxygen ≥ 60mmHg on room air or usual requirement level)

SECONDARY OUTCOMES:
Time to clinical stability | up to 2 weeks
  time to clinical stabilization
Early clinical stability rate | 3 days
  day 3 clinical stability rate
Late clinical stability rate | 7 days
  day 7 clinical stability rate
Hospital length of stay | 1 day (during hospital admission)
  length of hospital admission
Radiological improvement | 3 and 7 days
  improvement of lung infiltration or atelectasis
Broadening of antimicrobial spectrum | 1 day (during hospital admission)
  escalation antibiotics
Frequency of bronchoscopy for toileting | 1 day (during hospital admission)
  frequency of invasive lung care like bronchoscopy
In-hospital mortality | 1 day (during hospital admission)
  all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Eun Sun Kim, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No